CLINICAL TRIAL: NCT01443455
Title: Phase 2 Trial of Video Dance Versus Walking in Postmenopausal Sedentary Overweight Women
Brief Title: Adherence and Health Effects of Video Dance in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Stephanie Studenski, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO08080012; T32AG021885 (NIH); P30AG024827 (NIH)
Record Dates: First submitted 2011-09-27; First posted 2011-09-29 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Post Menopausal
Keywords: menopause; sedentary; overweight
MeSH Terms: conditions — Sedentary Behavior; Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- VideoDance (Experimental)
  Interventions: Behavioral: videodance
- Brisk Walking (Active Comparator)
  Interventions: Behavioral: Brisk Walking
- Delayed entry control (Other): Participants who are randomized to the delayed entry non-exercise control group receive the American Heart Association pamphlet, but no direct support for exercise implementation. After they have completed six months of follow up, they are invited to select any combination of dancing and walking that they prefer and then receive support and instruction according to the protocols described above.
  Interventions: Behavioral: delayed entry control

INTERVENTIONS:
Behavioral: videodance — Using a commercially available product called Dance Dance Revolution (DDR) this video-game based dancing system uses a game player, force sensing pad and software. The step sequences are set to a wide range of music and become more complex and frequent as the dancer gains skill. Participants are oriented over 2 weeks. For the rest of the first 3 months, the participant attends at least one supervised session per week. Participants may use the center for additional, unsupervised sessions and/or they can take a dance system home. They also receive brief behavioral intervention sessions for safety orientation, exercise education and adherence promotion. For the following 3 months, the participant enters the transition phase in which she is encouraged to continue to exercise but no formal supervision is provided.
  Other Names: Konami
  Arms: VideoDance
Behavioral: Brisk Walking — The overall goal is to increase the duration and speed of walking, using structure and supervision for the first three months, followed by reduced support in the second three months. For the first two weeks, each participant comes to the center at least twice a week to walk.They are encouraged to gradually increase effort and duration to a target of 150 minutes per week of brisk walking.Participants are taught to use Borg's ratings of perceived exertion and self-monitored heart rate to target their level of activity. The next 10 weeks include once weekly supervised sessions and additional sessions either at the center or in preferred community settings. The recommended goal is a minimum of 150 minutes per week of exercise in sessions of at least 10 -15 minutes duration.Participants are given pedometers in order to help them monitor their progress. After 12 weeks, the participant enters a transition phase for a further 3 months.
  Arms: Brisk Walking
Behavioral: delayed entry control — Participants who are randomized to the delayed entry non-exercise control group receive the American Heart Association pamphlet, but no direct support for exercise implementation. After they have completed six months of follow up, they are invited to select any combination of dancing and walking that they prefer and then receive support and instruction according to the protocols described above.
  --------------------------------------------------------------------------------
  Arms: Delayed entry control

SUMMARY:
This is a 6 month randomized clinical trial comparing video dance, brisk walking and delayed entry controls. The interventions have two phases; a 12 week initiation phase with substantial structure and supervision, followed by a 12 week transition phase, with reduced structure and supervision. Participants are 168 overweight or obese, sedentary postmenopausal women aged 50 to 65; 60 in each exercise arm and 48 in the wait list control group.

The following research questions will be assessed:

1. Is exercise adherence at 6 months better with video dance games compared to brisk walking?
2. Does video dance game exercise compared to wait list controls, induce beneficial changes in physical and mental health?
3. Does video dance game exercise compared to brisk walking better promote balance, attention and visual spatial skills, without loss of benefit to cardiovascular fitness?
4. Is video dance preferred to brisk walking for exercise among postmenopausal women? If so, who and why?

ELIGIBILITY:
Inclusion Criteria:

* Participants must be female
* age 50-65
* not currently exercising at least 20 minutes
* three times per week
* a BMI of 25 or higher

Exclusion Criteria:

* Exclusions are largely related to medical safety and include history of osteoporosis, osteoporotic fractures, active cardiovascular disease, uncontrolled hypertension, weight bearing pain that would limit exercise, seizure disorder or any medical condition or medication that would limit the safety of the study.

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2012-07-31 (Actual); Study Completion 2012-09-30 (Actual)

PRIMARY OUTCOMES:
Adherence | six months after randomization
  minutes per week of moderate or greater physical exercise activity assessed using accelerometers and activity diaries

SECONDARY OUTCOMES:
Endurance | 3 and 6 months
  timed 2 km walk
body composition | 6 months
  Lunar Prodigy DXA scanner for lean body mass and total fat mass
vascular health | 6 months
  blood pressure, pulse, lipid levels, fasting glucose, fasting insulin and C reactive protein
balance | 3 and 6 months
  timed one foot stand and timed narrow walk
personality | baseline
  NEO Personality Inventory
sleep quality | 3 and 6 monhts
  Pittsburgh Sleep Quality Index
visuospatial/constructional function | 3 and 6 monhts
  domain of the Repeatable Battery for the Assessment of Neuropsychological Status
attention domain | 3 and 6 monhts
  subtests of the Repeatable Battery for the Assessment of Neuropsychological Status
Useful Field of View | 3 and 6 monhts
  Useful Field of View test
step reaction time | 3 and 6 months
  Step Reaction Tasks

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie A Studenski, MD MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Jovancevic J, Rosano C, Perera S, Erickson KI, Studenski S. A protocol for a randomized clinical trial of interactive video dance: potential for effects on cognitive function. BMC Geriatr. 2012 Jun 6;12:23. doi: 10.1186/1471-2318-12-23. PMID 22672287